CLINICAL TRIAL: NCT03652584
Title: A Randomised Controlled Intervention Study Investigating the Effects of High Protein Diet on Body Composition, Strength, and Physical Performance in Postmenopausal Women
Brief Title: Effects of High Protein Diet on Muscle Mass, Strength, and Physical Performance in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Brazilian National Institute of Hormones and Women's Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 170019
Record Dates: First submitted 2018-08-17; First posted 2018-08-29 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Muscle Loss; Physical Disability
Keywords: postmenopause; diet; Skeletal muscle mass
MeSH Terms: conditions — Muscular Atrophy | interventions — Diet, High-Protein

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Protein Diet (Experimental): Low glycemic index dietary plan with 1.6 g/kg/day of protein for 6 months
  Interventions: Other: High Protein Diet
- Control Diet (Active Comparator): Low glycemic index dietary plan with 0.8 g/kg/day of protein for 6 months
  Interventions: Other: Control Diet

INTERVENTIONS:
Other: High Protein Diet
  Arms: High Protein Diet
Other: Control Diet
  Arms: Control Diet

SUMMARY:
Despite the importance of preventing muscle mass loss during senescence, only a few studies have investigated the relationship between diet and muscle mass in postmenopausal women. Therefore, the aim of this study is to investigate whether controlled protein consumption at the current Recommended Daily Allowance (RDA = 0.8 g/kg body weight) or twice the RDA (1.6 g/kg body weight) affects skeletal muscle mass, strength, and physical performance in postmenopausal women. In this parallel-group trial, participants were randomized for 6 months to low glycemic index diets with controlled protein consumption at the current RDA or twice the RDA, aimed to balance energy needs.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* Without mobility aids, able to perform activities of daily living independently

Exclusion Criteria:

* Use of hormone therapy in the past 3 months
* Insulin therapy
* Previous diagnosis of heart disease
* Untreated thyroid diseases
* Conditions affecting neuromuscular function

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change in whole-body and appendicular lean mass | 6 months
  measured by dual-energy X-ray absorptiometry

SECONDARY OUTCOMES:
Change in isometric hand grip strength | 6 months
  measured by dynamometry
Change in usual gait speed | 6 months
  in a 4-m course
Change in systolic blood pressure | 6 months
  in mmHg
Change in diastolic blood pressure | 6 months
  in mmHg
Change in fat mass | 6 months
  measured by dual-energy X-ray absorptiometry
Change in resting metabolic rate | 6 months
  measured by indirect calorimetry
Change in total cholesterol, high-density lipoprotein cholesterol, and triglycerides | 6 months
  determined by colorimetric-enzymatic methods
Change in glucose | 6 months
  determined by the hexokinase method
Change in insulin | 6 months
  measured by chemiluminescence immunoassays
Change in high-sensitivity C-reactive protein | 6 months
  measured by nephelometric method

CONTACTS AND LOCATIONS:
Overall Officials: Poli Mara Spritzer, MD PhD, Study Director — Federal University of Rio Grande do Sul